CLINICAL TRIAL: NCT01571583
Title: Open-Label, Phase 3b Study To Determine Efficacy and Safety of Telaprevir, Pegylated-Interferon-alfa-2a and Ribavirin in Hepatitis C Genotype 1 Infected, Stable Liver Transplant Subjects
Brief Title: An Efficacy and Safety Study of Telaprevir in Patients With Genotype 1 Hepatitis C Infection After Liver Transplantation
Acronym: REPLACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018721; VX-950HPC3006 (Other: Janssen-Cilag International NV, Belgium); 2011-004724-35 (EudraCT Number)
Record Dates: First submitted 2011-12-16; First posted 2012-04-05 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Hepatitis C Virus (HCV) Infection
Keywords: Chronic HCV infection; Genotype 1 chronic HCV; Liver transplantation; Hepatitis C; Hep C; HCV; Telaprevir; Pegylated-Interferon-alfa-2a; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Infections | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telaprevir+Peg-IFN-alfa-2a+Ribavirin (Experimental): Patients will be treated for 12 weeks with telaprevir in combination with Pegylated interferon alfa-2a (Peg-IFN-alfa-2a) and ribavirin followed by 36 weeks of treatment with Peg-IFN-alfa-2a and ribavirin alone.
  Interventions: Drug: Telaprevir; Drug: Pegylated interferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir — Type=exact number, unit=mg, number=375, form=tablet, route=oral. Patients will receive 2 oral tablets (750 mg) every 8 hours for 12 weeks.
Drug: Pegylated interferon alfa-2a — Type=exact number, unit=µg, number=180, form=injection, route=subcutaneous. 180 microgram (µg) per week, subcutaneous injection, for 48 weeks.
Drug: Ribavirin — Type=exact number, unit=mg, number=200, form=tablet, route=oral. Starting from 600 mg (3 tablets) per day on Day 1. This dose will become higher or lower based on blood results and the investigators opinion (to a goal of 1000 to 1200 mg/day [5 to 6 tablets] based on subject weight), twice daily regimen, for 48 weeks.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of telaprevir in combination with Peg-IFN-alfa-2a and ribavirin in stable liver transplant patients with chronic hepatitis C virus (HCV) genotype 1.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter study in genotype 1 chronic HCV infected liver transplant patients who will be treated for 12 weeks with telaprevir 750 mg every 8 hours given in combination with Peg-IFN-alfa-2a and ribavirin followed by 36 weeks of treatment with Peg-IFN-alfa-2a and ribavirin alone. The total treatment duration will be 48 weeks. Safety will be evaluated throughout the study and will include evaluations of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* First time liver transplant recipient whose primary pre-transplant diagnosis was chronic hepatitis C genotype 1
* More than 6 months to 10 years post-liver transplant
* Patient did or did not receive treatment for HCV prior to liver transplantation
* Patient must agree to have a liver graft biopsy during the screening period unless they had a biopsy within three months of the screening period (for patients between 6 months and one year post transplant) or within six months of the screening period (for patients who are more than one year post transplant)
* A female patient of childbearing potential and a nonvasectomized male patient who has a female partner of childbearing potential must agree to the use of 2 effective methods of birth control from screening until 6 months (female patient) or 7 months (male patient) after the last dose of ribavirin

Exclusion Criteria:

* Patient is currently infected or co-infected with HCV of another genotype than genotype 1
* Patient received treatment for hepatitis C following liver transplantation
* Patient has history of decompensated liver disease or shows evidence of significant liver disease in addition to hepatitis C
* Patient with human immunodeficiency virus or hepatitis B virus co-infection
* Patient with active malignant disease or history of malignant disease within the past 5 years (with the exception of treated basal cell carcinoma or hepatocellular carcinoma)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving sustained virologic response (SVR) 12 planned | Week 60
  SVR12 planned is defined as having plasma hepatitis C virus (HCV ) ribonucleic acid (RNA) level less than 25 IU/mL 12 weeks after the last planned dose of study medication.

SECONDARY OUTCOMES:
Number of patients achieving SVR12 planned(c) | Week 60
  SVR12 planned(c) is defined as having undetectable plasma HCV RNA levels 12 weeks after the last planned dose of study drugs.
Number of patients achieving SVR24 planned | Week 72
  SVR24 planned is defined as having plasma HCV RNA levels less than 25 IU/mL 24 weeks after the last planned dose of study medication.
Number of patients achieving SVR24 planned(c) | Week 72
  SVR24 planned(c) is defined as having an undetectable plasma HCV RNA level 24 weeks after the last planned dose of study medication.
Number of patients having an undetectable HCV RNA level at Week 4 of treatment | Week 4
Number of patients having an undetectable HCV RNA level at Week 12 of treatment | Week 12
Number of patients having undetectable HCV RNA levels at Week 4 and Week 12 of treatment | Week 4 and Week 12
Number of patients having an undetectable HCV RNA level at the actual end of treatment | Week 48
Number of patients having an undetectable HCV RNA level at the planned end of treatment | Week 48
Number of patients having less than 25 IU/mL at the planned end of treatment | Week 48
Number of patients with on-treatment virologic failure | Week 48
  Virologic failure is defined as patients who meet a virologic stopping rule and/or meet the definition of viral breakthrough.
Number of patients with relapse after undetectable HCV RNA at actual end of treatment | Week 48
  Number of patients who relapse, defined as having confirmed detectable HCV RNA during the follow-up period after previous undetectable HCV RNA (less than 25 IU/mL, target not detected) at actual end of treatment.
Number of patients with relapse after undetectable HCV RNA at planned end of treatment | Week 48
  Number of patients who relapse, defined as having confirmed detectable HCV RNA during the follow-up period after previous undetectable HCV RNA (less than 25 IU/mL, target not detected) at planned end of treatment.
Number of patients with relapse after previous HCV RNA less than 25 IU/mL at planned end of treatment | Week 48
  Number of patients who relapse, defined as having confirmed detectable HCV RNA during the follow-up period after previous HCV RNA less than 25 IU/mL at planned end of treatment.
Number of patients with viral breakthrough | Week 48
  Number of patients with viral breakthrough (defined as an increase more than 1 log in HCV RNA level from the lowest level reached, or a value of HCV RNA more than 100 IU/mL in patients whose HCV RNA has previously become less than 25 IU/mL during treatment).
Change from baseline in log HCV RNA values | Up to Week 52
  Change from baseline in log HCV RNA values at each time point during treatment.
Number of patients who have changes in liver graft biopsy histology | Up to Week 72
Number of patients with adverse events | Up to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV, Belgium Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (21):
- Austria (2):
  - Linz
  - Vienna
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Liège
- France (5):
  - Clichy
  - Marseille
  - Montpellier
  - Rennes Cedex N/A
  - Villejuif
- Germany (5):
  - Essen
  - Frankfurt A. M.
  - Hanover
  - Leipzig
  - Münster
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia
- United Kingdom (2):
  - Birmingham
  - London

REFERENCES:
- See also: Open-Label, Phase 3b Study To Determine Efficacy and Safety of Telaprevir, Pegylated-Interferon-alfa-2a and Ribavirin in Hepatitis C Genotype 1 Infected, Stable Liver Transplant Subjects(18137). — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3339&filename=20150616_VX-950HPC3006(CR018721)_PRF.pdf